CLINICAL TRIAL: NCT06284161
Title: Contribution of the Combined Quadriceps Test (QCT) in the Diagnosis, Mechanistic Understanding and Follow-up of Amyotrophic Lateral Sclerosis
Brief Title: QCT in ALS Diagnosis, Mechanistic Understanding and Follow-up
Acronym: PEM-SLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2020 GUY; 2020-A02765-34 (Other: ANSM)
Record Dates: First submitted 2022-06-21; First posted 2024-02-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Quadriceps Combined Test; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Evoked Potentials, Motor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quadriceps Combined Test (Other)
  Interventions: Diagnostic Test: Quadriceps Combined Test

INTERVENTIONS:
Diagnostic Test: Quadriceps Combined Test — The recording of the motor response on the quadriceps is done using self-adhesive surface electrodes on the motor point of the vastus medialis muscles (active electrodes) and on the patella (reference electrode), using a classic electromyography device that allows calculations and measurements of amplitude, duration and speed.
  Other Names: Motor- Evoked Potentials

SUMMARY:
Multidisciplinary management of amyotrophic lateral sclerosis (ALS) can significantly increase survival but also improve the quality of life of patients. The evaluation of cortical-spinal motor neuron damage is currently based only on the assessment of clinical data. However, the alteration of the central motor pathway and conduction can be identified and quantified by different techniques using motor-evoked potentials (MEP). The combined quadriceps test (QCT) has been developed to assess central and peripheral motor pathway conduction. This test allows to quantify central and peripheral part of a mixed disorder, and to detect physiological hyporeflexia or hyperreflexia which, in the case of suspected ALS, can lead to interpretation problems.

The evolution of the QCT parameters during the course of pathology will lead to determine the preponderance of an initial central involvement, but also its extension throughout the pathology. The study of these parameters as well as the clinical course of the disease could reveal a correlation between peripheral and central involvement. This link would provide arguments in favor of pathophysiological hypotheses of disease onset and progression. From a prognostic point of view and depending on the quantification of central and peripheral involvement, the QCT would make it possible to characterize the different ALS phenotypes. This phenotypic characterization would help identify prognostic factors at diagnosis.

The investigators propose a cohort study with the exploration of central motor neuron damage by QCT during the course of ALS in order to provide arguments for a better mechanistic understanding and follow-up of this disease with a poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

* A male or female patient of legal age with suspected ALS (bulbar or spinal) who meets the criteria for "possible", "probable" or "definite" ALS according to the Awaji criteria
* Able to give informed consent to participate in the research
* Enrolled in a Social Security plan

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Severe progressive pathology other than ALS.
* Comorbidities with another neurological disease altering motor skills.
* Contraindication to trans-cranial magnetic stimulation: epilepsy, pacemaker, intracranial ferromagnetic foreign body (clip, aneurysm, implants)...
* Chronic alcoholism
* Cognitive disorders or major incapacity making it impossible to understand the study and sign an informed consent (fronto-temporal dementia, psychiatric conditions of psychotic type, language disorders)
* Refusal to participate.
* Patients under legal protection (guardianship, curators, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Parameters from the QCT (Quadriceps Combined Test) | At inclusion
  Measure of amplitude of M
Parameters from the QCT (Quadriceps Combined Test) | Month 6
  Measure of amplitude of M
Parameters from the QCT (Quadriceps Combined Test) | Month 12
  Measure of amplitude of M
Parameters from the QCT (Quadriceps Combined Test) | month 18
  Measure of amplitude of M
Parameters from the QCT (Quadriceps Combined Test) | month 24
  Measure of amplitude of M
Parameters from the QCT (Quadriceps Combined Test) | At inclusion
  measure of TCP response,
Parameters from the QCT (Quadriceps Combined Test) | month 6
  measure of TCP response,
Parameters from the QCT (Quadriceps Combined Test) | month 12
  measure of TCP response,
Parameters from the QCT (Quadriceps Combined Test) | month 18
  measure of TCP response,
Parameters from the QCT (Quadriceps Combined Test) | month 24
  measure of TCP response,
Parameters from the QCT (Quadriceps Combined Test) | At inclusion
  measure of TCC response
Parameters from the QCT (Quadriceps Combined Test) | month 6
  measure of TCC response
Parameters from the QCT (Quadriceps Combined Test) | month 12
  measure of TCC response
Parameters from the QCT (Quadriceps Combined Test) | month 18
  measure of TCC response
Parameters from the QCT (Quadriceps Combined Test) | month 24
  measure of TCC response
Parameters from the QCT (Quadriceps Combined Test) | At inclusion
  ratio calculation of amplitude
Parameters from the QCT (Quadriceps Combined Test) | month 6
  ratio calculation of amplitude
Parameters from the QCT (Quadriceps Combined Test) | month 12
  ratio calculation of amplitude
Parameters from the QCT (Quadriceps Combined Test) | month 18
  ratio calculation of amplitude
Parameters from the QCT (Quadriceps Combined Test) | month 24
  ratio calculation of amplitude
Parameters from the QCT (Quadriceps Combined Test) | At inclusion
  ratio calculation of T/MEP latency ratio
Parameters from the QCT (Quadriceps Combined Test) | month 6
  ratio calculation of T/MEP latency ratio
Parameters from the QCT (Quadriceps Combined Test) | month 12
  ratio calculation of T/MEP latency ratio
Parameters from the QCT (Quadriceps Combined Test) | month 18
  ratio calculation of T/MEP latency ratio
Parameters from the QCT (Quadriceps Combined Test) | month 24
  ratio calculation of T/MEP latency ratio
Parameters from the QCT (Quadriceps Combined Test) | At inclusion
  ratio calculation of T/MEP amplitude ratio.
Parameters from the QCT (Quadriceps Combined Test) | month 6
  ratio calculation of T/MEP amplitude ratio.
Parameters from the QCT (Quadriceps Combined Test) | month 12
  ratio calculation of T/MEP amplitude ratio.
Parameters from the QCT (Quadriceps Combined Test) | month 18
  ratio calculation of T/MEP amplitude ratio.
Parameters from the QCT (Quadriceps Combined Test) | month 24
  ratio calculation of T/MEP amplitude ratio.

SECONDARY OUTCOMES:
Clinical and paraclinical likely course data | At inclusion
  MRC (Medical Research Council) scale for the evaluation of muscular strength. Score from 0 to 5. Higher score means normal movement
Clinical and paraclinical likely course data | At inclusion
  ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating) scale score. Score from 0 to 48.
Clinical and paraclinical likely course data | At inclusion
  Spirometry data : Slow Vital Capacity
Clinical and paraclinical likely course data | At inclusion
  Spirometry data : Maximal Inspiratory Pressure
Clinical and paraclinical likely course data | At inclusion
  Spirometry data : Maximal Exhalation Pressure
Clinical and paraclinical likely course data | At inclusion
  Weight
Clinical and paraclinical likely course data | At inclusion
  Percentage of weight loss
Clinical and paraclinical likely course data | At inclusion
  Oxymetry
Clinical and paraclinical likely course data | At inclusion
  Non-Invasive Ventilation implementation (yes or no)
Clinical and paraclinical likely course data | At inclusion
  Gastrostomy implementation (yes or no)
Clinical and paraclinical likely course data | At inclusion
  Survival
Clinical and paraclinical likely course data | Every 3 months up to 2 years
  MRC (Medical Research Council) scale for the evaluation of muscular strength. Score from 0 to 5. Higher score means normal movement
Clinical and paraclinical likely course data | Every 3 months up to 2 years
  ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating) scale score. Score from 0 to 48.
Clinical and paraclinical likely course data | Every 3 months up to 2 years
  Spirometry data : Slow Vital Capacity
Clinical and paraclinical likely course data | Every 3 months up to 2 years
  Spirometry data : Maximal Inspiratory Pressure
Clinical and paraclinical likely course data | Every 3 months up to 2 years
  Spirometry data : Maximal Exhalation Pressure
Clinical and paraclinical likely course data | Every 3 months up to 2 years
  Weight
Clinical and paraclinical likely course data | Every 3 months up to 2 years
  Percentage of weight loss
Clinical and paraclinical likely course data | Every 3 months up to 2 years
  Oximetry
Clinical and paraclinical likely course data | Every 3 months up to 2 years
  Non-Invasive Ventilation Implementation (yes or no)
Clinical and paraclinical likely course data | Every 3 months up to 2 years
  Gastrostomy implementation (yes or no)
Clinical and paraclinical likely course data | Every 3 months up to 2 years
  Survival

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Guy, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France